CLINICAL TRIAL: NCT06953245
Title: Collecting Patient-Reported Experiences With Radiation Dermatitis in Breast Cancer Patients Undergoing Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR2431; NCI-2025-01198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-007996 (Other: Mayo Clinic Institutional Review Board); ROR2431 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete a survey on study, completed as a brief interview.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates patient-reported experiences of radiation dermatitis in patients with breast cancer undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18
* Patients diagnosed with breast cancer
* Currently undergoing or recently completed radiotherapy
* Willing to provide verbal/oral consent

Exclusion Criteria:

* Persons < 18
* Inability to provide verbal consent
* Non-English speakers (unless translations are available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer who are currently undergoing or recently completed radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient experiences with radiation dermatitis | Baseline (at enrollment)
  Themes will be collected during a brief interview following agreement to participate. Common themes related to physical, emotional, and social impacts of radiation dermatitis will be categorized and quantified to provide a comprehensive understanding of the patient experience.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S. Corbin, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials